CLINICAL TRIAL: NCT00005060
Title: A Phase III Trial of Preoperative vs. Postoperative Chemotherapy With Taxotere-Cisplatin-5FU (TCF) in Patients With Locally Advanced Operable Gastric Carcinoma
Brief Title: Combination Chemotherapy and Surgery in Treating Patients With Locally Advanced Stomach Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 43/99; SWS-SAKK-43/99 (Other: SAKK); EU-99042
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Gastric Cancer
Keywords: stage II gastric cancer; stage III gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Taxotere-Cisplatin-5FU preoperatively (Active Comparator): TCF preoperatively
  Interventions: Drug: Taxotere-Cisplatin-5FU
- Immediate surgery followed by TCF (Active Comparator): Surgery followed by Taxotere-Cisplatin-5FU
  Interventions: Drug: Immediate surgery

INTERVENTIONS:
Drug: Taxotere-Cisplatin-5FU — Preoperatively
  Arms: Taxotere-Cisplatin-5FU preoperatively
Drug: Immediate surgery — Immediate surgery followed by Taxotere-Cisplatin-5FU
  Arms: Immediate surgery followed by TCF

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug with surgery may kill more tumor cells. It is not yet known if chemotherapy followed by surgery is more effective than surgery followed by chemotherapy for stomach cancer.

PURPOSE: This randomized phase III trial is studying surgery followed by combination chemotherapy to see how well it works compared to combination chemotherapy followed by surgery in treating patients with locally advanced stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare, by intention to treat analysis, feasibility and efficacy of 4 courses of docetaxel, cisplatin, and fluorouracil as preoperative or postoperative chemotherapy in patients with locally advanced operable gastric carcinoma.
* Evaluate the predictive values of some biological and molecular tumor parameters on response to chemotherapy, metastasis and survival in this patient population.

OUTLINE: This is a randomized, open label, multicenter study. Patients are stratified according to study center, tumor site (affecting the Z-line (cardia carcinoma Siewart II and III) vs rest of the stomach), and nodal status (positive vs negative). Patients are randomized to either preoperative chemotherapy followed by surgery (arm I) or surgery followed by postoperative chemotherapy (arm II).

* Arm I: Patients receive docetaxel IV over 1 hour followed by cisplatin IV over 4 hours on day 1, and fluorouracil IV continuously on days 1-14 every 3 weeks. Patients are evaluated after 2 courses and patients with progressive disease proceed to immediate surgery. Otherwise, treatment continues for a total of 4 courses in the absence of unacceptable toxicity or disease progression. Between 3-5 weeks following day 1 of the last course of chemotherapy, patients undergo gastric resection.
* Arm II: Patients undergo immediate gastric resection. Beginning 3-6 weeks after surgery, patients receive 4 courses of docetaxel, cisplatin, and fluorouracil as in arm I.

Quality of life is assessed before the first and third courses of chemotherapy, before and after surgery, and then at 1, 3, and 6 months.

Patients are followed every 3 months for 3 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 240 patients (120 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed locally advanced gastric carcinoma that is considered operable

  * T3-4, Nx, M0 OR
  * Tx, N+, M0
* Lymph nodes considered positive by sonography should be at least 2 of the following:

  * Round
  * Echopoor
  * Sharp borders
  * At least 0.5 cm
* No distant metastases, including peritoneal carcinomatosis

  * CT scan and peritoneal lavage mandatory

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* 0-2

Life expectancy:

* Greater than 12 weeks

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* AST or ALT no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Adequate renal function within limits to allow for treatment with cisplatin

Cardiovascular:

* No unstable cardiac disease requiring treatment
* No congestive heart failure or angina pectoris even if medically controlled
* No significant arrhythmias
* No myocardial infarction within past 6 months
* Ejection fraction greater than 50% on cardiac sonography or MUGA scan

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior malignancy except basal cell carcinoma of the skin or adequately treated carcinoma in situ of the cervix
* No grade 2 or greater peripheral neuropathy of any origin (e.g., alcohol, diabetic)
* No history of anaphylaxis
* No other serious concurrent illness or medical condition that would preclude study therapy
* No history of significant neurologic or psychiatric disorders (e.g., psychotic disorders, dementia, or seizures)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent biologic therapy for gastric carcinoma

Chemotherapy:

* No other concurrent chemotherapy for gastric carcinoma

Endocrine therapy:

* No concurrent endocrine therapy for gastric carcinoma

Radiotherapy:

* No concurrent radiotherapy for gastric carcinoma

Surgery:

* See Disease Characteristics

Other:

* At least 30 days since prior treatment in a clinical trial
* No other concurrent experimental drugs
* No other concurrent anticancer therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 1999-11; Primary Completion 2005-11 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Event-free survival

SECONDARY OUTCOMES:
Overall survival
Time to treatment failure measured after completion of study treatment
Toxicity measured after completion of study treatment
Rate of complete resection (RO) and postoperative mortality as measured after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Morant, MD, Study Chair — Tumor Zentrum ZeTup St. Gallen und Chur
Locations (3):
- European Institute of Oncology, Milan, Italy
- Switzerland (2):
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Zentrum fuer Tumordiagnostikund Praevention, Sankt Gallen